CLINICAL TRIAL: NCT00043433
Title: Study of T900607-Sodium in Chemotherapy Naive Patients With Hepatocellular Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tularik (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-607-004
Record Dates: First submitted 2002-08-08; First posted 2002-08-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

INTERVENTIONS:
Drug: intravenous T900607-sodium

SUMMARY:
The purpose of the study is to determine whether T900607-sodium is effective and safe in treating hepatocellular carcinoma, a type of liver cancer.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of HCC
* Child-Pugh liver classification of A or B
* Subjects must not have received prior chemotherapy or radiotherapy for their HCC
* At least 18 years of age
* Bidimensionally measurable disease amenable to CT scanning. At least one lesion must be least 1 X 1 cm in size.
* Karnofsky performance status of at least 70%
* Estimated life expectancy of at least 12 weeks
* Females of childbearing potential must have a negative pregnancy test and agree to use an effective contraceptive
* Subject must be able to comply with study procedures and follow-up examinations.
* Signed written informed consent
* Lab Values (obtained ≤ 7 days prior to study enrollment):
* ANC at least 1.5x10e9/L,
* Platelet count at least 100x10e9/L,
* Creatinine within 2 times upper limit of normal
* AST and ALT within 5 times upper limit of normal
* Bilirubin within 1.5 times upper limit of normal
* Albumin great than 2.8 g/dL

Exclusion Criteria

* Severe, concurrent disease, infection or co-morbidity that, in the judgment of the investigator, would make the subject inappropriate for enrollment
* NYHA Class III/IV cardiac disease, left ventricular ejection fraction (LVEF) of <50%, or acute anginal symptoms
* Patients who have received any investigational agent within 4 weeks of enrollment
* Patients who are pregnant or breast-feeding
* History of prior malignancy other than cancer studied within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* History of central nervous system metastases or carcinomatous meningitis
* Major surgery within 4 weeks of enrollment
* Patients who have received prior chemotherapy, chemoembolization, immunotherapy, or radiotherapy for their HCC. Prior surgical resection, intratumoral ethanol injection, hormonal therapy, cryosurgery, radiofrequency ablation, selective internal radiation or embolization, is permitted ONLY if > 6 weeks has passed since therapy and there is an indicator lesion (> 1 x 1 cm) outside the area of prior treatment (recurrence at the margin or resection is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Charlene Sum, Study Chair — Tularik
Locations (12):
- United States (11):
  - Scripps Health Center, La Jolla, California
  - University of California San Diego, La Jolla, California
  - George Washington University, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Queen Mary Hospital, Hong Kong, China